CLINICAL TRIAL: NCT02842645
Title: Growth-Health and Development in Children Exposed to Drugs During Pregnancy.
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/3301
Record Dates: First submitted 2011-04-01; First posted 2016-07-25 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Growth Failure; Mental Health Disorder; Foetal Exposure During Pregnancy
Keywords: Foetal Exposure During Pregnancy; Health; Growth
MeSH Terms: conditions — Failure to Thrive; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Children born at term and not exposed to drugs during pregnancy
- Case: Case = Children exposed to drugs during pregnancy

SUMMARY:
"Children exposed to alcohol or drugs during pregnancy: Growth, health and development" Background Children exposed to drugs during pregnancy are at risk of developmental disorders. The scope and size of this problem is poorly known in Norway.

Alcohol has a known teratogenic effect on the fetus. How other drugs affect the fetus, is associated with more uncertainty. Withdrawal in the neonatal period has been perceived as the main problem. There is less knowledge about long-term outcome of exposure to drugs during pregnancy.

Aim The aim of the study is to investigate the physical and mental health of children exposed to drugs during pregnancy. Identify the children's need for measures in the home and school, and how many of the children who are taken care of in fostercare.

A sample of the children will be offered radiological examination of the brain (f-MRI). The purpose is to study the relationship between exposure to drugs, child development, environment and organic brain dysfunction.

Design The project is a quantitative study. The relationship between exposure to drugs and development will be measured by questionnaires, clinical examination, neuropsychological tests and radiological examination (f-MRI).

Children aged 2-15years who were referred, examined or treated for drug related problems at the Department of Pediatrics, Haukeland University Hospital will be invited to participate in the study.

Information retrieval and examination of the children are expected to be completed during 2011. Data analysis and further processing of data are expected to be completed during 2013.

ELIGIBILITY:
Inclusion Criteria:

* Foetal exposure of drugs during pregnancy.

Exclusion Criteria:

* Non exposed children

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children exposed to drugs during pregnancy are followed up at school age regarding mental disorders and status of their care situation.
  Approximately 130 children are invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mental Health Disorder | 2012
  Questionaire regarding mental health: Strength and Difficulties Questionnaires

OTHER OUTCOMES:
Social status | 2012
  Questionaire regarding social status

CONTACTS AND LOCATIONS:
Overall Officials: Irene B Elgen, Professor, Principal Investigator — Department of Child and Adolscent Psychiatry, Haukeland University Hospital, N-5018 Bergen
Locations (2):
- Norway (2):
  - Haukeland universitet sykehus, Bergen
  - Haukelans universitetssykehus, Bergen

IPD SHARING:
Plan to Share IPD: No